CLINICAL TRIAL: NCT06616558
Title: A Single-Center, Open-Label, Randomized Clinical Study to Evaluate the Oil Control Efficacy, Moisture Assessment and Skin Barrier Integrity of an Investigational Product in Adult Participants With Oily Facial Skin
Brief Title: A Study to Assess the Effectiveness of Sunscreen on Oil Control, Moisturization, and Skin Barrier Integrity in Adults With Oily Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JNTL Consumer Health (Brasil) LTDA (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CS2024SK100142
Record Dates: First submitted 2024-08-13; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-06

CONDITIONS: Oily Skin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sunscreen Home Usage (Experimental): Participants will use the Sunscreen in normal conditions at home for 28 +/- 2 days, returning to the Site after 7 days of product use, then make the last study visit to complete the final analysis.
  Interventions: Other: Sunscreen SPF 70
- Oil Control Assessment Product Application (Experimental): An amount of Investigational Product will be topically applied to malar and forehead areas (after cleansing the face) on one randomized side of the participant's face by a qualified technician to perform the assessment of a 12-hour kinetics. After the evaluations the product will be removed.
  Interventions: Other: Sunscreen SPF 70
- Oil control Assessment (Control) (No Intervention): On the randomized half-side (malar and forehead areas), no product will be applied and this will be the control for evaluating the product's oil control during the 12-hour kinetics.

INTERVENTIONS:
Other: Sunscreen SPF 70 — Participants will topically apply sunscreen SPF 70
  Arms: Sunscreen Home Usage
Other: Sunscreen SPF 70 — On the randomized side of the half-face, the product will be applied by a qualified technician
  Arms: Oil Control Assessment Product Application

SUMMARY:
The purpose of this trial is to evaluate 1) the efficacy of an investigational product (sunscreen) when compared to a control area (without product application) in controlling oiliness, oil shine and the effect on pores appearance in a 12-hour kinetics through a) Instrumental measurements, b) Expert Grader and c) Perceived efficacy; 2) the efficacy of an investigational product in reducing oiliness, improving hydration, the pores appearance and the integrity of the skin barrier, after 7 days of use and after 28 ± 2 days of use through instrumental measurements and perceived efficacy questionnaires.

DETAILED DESCRIPTION:
The objectives of this study are:

To evaluate the efficacy of an investigational product (sunscreen) when compared to a control area (without product application) in controlling oiliness, oil shine and the effect on pores appearance in a 12-hour kinetics:

* Instrumental measurements with the Sebumeter® SM 815 equipment to assess oiliness control;
* Clinical efficacy evaluation carried out by Expert Grader
* Perceived efficacy through perception questionnaires

To evaluate the efficacy of an investigational product in reducing oiliness, improving hydration, pores appearance and the integrity of the skin barrier, after 7 days of use and after 28 ± 2 days of use, under normal conditions of use in adult participants through the following evaluations:

* Instrumental measurements with the Sebumeter® SM 815 equipment before and after 7 and 28 ± 2 days of use on the face to assess oil reduction;
* Instrumental measurements with the Corneometer® before and after 7 and 28 ± 2 days of use on the face to assess skin hydration;
* Instrumental measurements with the Tewameter® TM 300 before and after 7 and 28 ± 2 days of use on the face to assess the integrity/maintenance of the skin barrier;
* Facial images captured using Visia® CR equipment before and after 7 and 28 ± 2 days of use on the face;
* Perceived efficacy through perception questionnaires answered by research participants after 7 and 28 ± 2 days of use on the face;
* Open-ended emotional statement after 28 ± 2 days.

ELIGIBILITY:
Inclusion Criteria:

* Men and/or Women;
* 18 to 55 years old;
* Phototypes I to VI according to the Fitzpatrick classification;
* Subjects of any ethnicity according to Brazilian Institute of Geography and Statistics (IBGE) criteria
* Integral skin in the test areas;
* Subjects with oily skin, confirmed by instrumental measurements: (sebumetry value of at least 100μg/cm² in the frontal region (average of 3 measurements)).
* Subjects with face oil shine - confirmed by Dermatologist;
* Subjects with enlarged pores on the face - confirmed by a Dermatologist;
* Subjects with self-perceived combination/oily or very oily skin on the face;
* Subjects with a self-perceived oil shine on the face;
* Subjects with self-perceived enlarged pores on the face;
* Do not use cosmetic products (including usual soap) the night before the visit and do not wash your face after 10 p.m. the day before the visit;
* For male subjects: who agree to shave 48 hours before the visits;
* Generally, in good health based on medical history reported by the subject;
* Subjects able to read, write, speak, and understand Portuguese;
* Agreeing to adhere to the procedures and requirements of the study and attending the Site on the day(s) and time(s) set for the evaluations;
* Subjects who signed the terms Informed Consent Document (ICD) and Informed Consent Image Disclosure (ICID);
* Intends to complete the study and is willing and able to follow all the study instructions.

Exclusion Criteria:

* Has known allergies or adverse reactions to common topical skin care products including sunscreens;
* Presents a skin condition that may confound the study results (specifically psoriasis, eczema, atopic dermatitis, cutaneous xerosis, erythema, or active skin cancer);
* Have primary/secondary lesions (e.g. scars, ulcers, vesicles) or tattoos in the test areas;
* Has self-reported Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication;
* Is taking a medication that would mask an Adverse Event (AE) or confound the study results, including:

  * Immunosuppressive or steroidal drugs within 2 months before Visit 1*
  * Non-steroidal anti-inflammatory drugs within 5 days before Visit 1* (For Oxaprozin and Piroxicam consider 2 weeks before visit 1).
  * Antihistamines within 2 weeks before Visit 1* *If an individual is taking one of these medication types, the individual is not considered eligible at screening. However, if a subject begins using one of these medications during the study, the Study Physician should be consulted to consider the impact of the specific medication on subject safety and/or the study results, as described in section "Concurrent/Concomitant Medication".
* Use of any other products capable of interfering with the study evaluations, at the discretion of the dermatologist;
* Subjects who have undergone invasive aesthetic or dermatological treatment in the test area within 2 months prior to the start of the study or during the study;
* Subjects who had used cosmetic products to treat oiliness/shine on the same area (face) within 14 days prior to the start of the study;
* Subjects who are using any medication to treat diseases of the face or eyes;
* Subjects who reported being pregnant, or planning to become pregnant during the study;
* Has a history of or a concurrent health condition/situation which may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study;
* Simultaneously taking part in another study;
* Being an employee/contractor or close relative of the Principal Investigator, Study Site, or Sponsor;
* Excessive hair in the assessment area that could interfere with instrumental measurements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | Up to 28 days
  Number of participants with adverse events will be reported. An adverse event is any untoward medical occurrence in a clinical study participant temporally associated with the clinical investigation, whether or not the event has a causal relationship to the participants' participation in the trial. It is therefore any unfavorable and unintended sign (including an abnormal finding), symptom, or disease that occurs during the trial. This can include any occurrence that is new in onset, an aggravation of severity/frequency of a baseline condition, or abnormal results of diagnostic procedures, including laboratory test abnormalities.
Change From Baseline in Skin Oil Control Assessment During 12-hour Kinetics | Day 1: Baseline, 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours and 12 hours
  Change from baseline in skin oil control will be reported. The facial oil control will be assessed by a trained technician using instrumental measurements with the Sebumeter SM 815. The Sebumeter measures amount of sebum per area.
  Sebumetric measurements will be taken in the forehead region of each half of the face during a 12-hour kinetics. One half of the forehead region will contain the Investigational Product and the other half will be the control, with no product applied.
Participant's Self-perceived Questionnaire to Assess the Clinical Effectiveness of the Sunscreen During 12-hour Kinetics | Day 1: Baseline, 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours and 12 hours
  Participant's self-perceived questionnaire to assess the clinical effectiveness of the sunscreen on oil and shine control. Participants will answer 6 questions and rate as: totally disagree, disagree, neither agree nor disagree, agree and totally agree. The area to be evaluated is half face with and without product applied.
Change From Baseline in Clinical Effectiveness on Oil Shine | Day 1: Baseline, 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours and 12 hours
  Change from Baseline in Clinical Effectiveness Assessment on Oil Shine will be reported. A 10-point ordinal scale (0 to 9) will be used. Therefore, as it is an ordinal scale, the intermediate points do not have an established definition. The evaluated area will be each half face and the scale to be used is defined from 0 = Dull, matte skin to 9 = Very intense oil shine, very oily skin. The time-points will me compared in terms of statistical improvement (improvement of oiliness shine (regulation)) versus the baseline.
Change From Baseline in Clinical Effectiveness on Pores Appearance | Day 1: Baseline, 30 minutes, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours and 12 hours
  Change from Baseline in Clinical Effectiveness Assessment on Pores Appearance will be reported. A 10-point ordinal scale (0 to 9) will be used. Therefore, as it is an ordinal scale, the intermediate points do not have an established definition. The evaluated area will be each half face and the scale to be used is defined from 0 =small, hardly visible to 9 = large, easily visible. The time-points will me compared in terms of statistical improvement (improvement in the appearance (number and/or size) of pores) versus the baseline.
Change From Baseline in Skin Oil Control Assessment | Baseline (Day 1), Day 7 and Day 28 +/- 2 days
  Change from baseline in skin oil control will be reported. The facial oil control will be assessed by a trained technician using instrumental measurements with the Sebumeter SM 815. The Sebumeter measures amount of sebum per area. Sebumetric measurements will be taken in the forehead region.
Change From Baseline in Skin Barrier Integrity | Baseline (Day 1), Day 7 and Day 28 +/- 2 days
  Change from baseline in skin barrier integrity will be reported. The facial skin barrier will be assessed by a trained technician using instrumental measurements with the Tewameter TM 300. The Tewameter measures transepidermal water loss (TEWL) that is the flow of water out of the skin. TEWL measurement will be taken in the nasolabial region of one randomized half of the face.
Change From Baseline in Skin Hydration | Baseline (Day 1), Day 7 and Day 28 +/- 2 days
  Change from baseline in skin hydration will be reported. The facial skin hydration will be assessed by a trained technician using instrumental measurements with the Corneometer® CM825. The Corneometer measures the dielectric constant of the skin. The dielectric constant of skin will change with water content of the stratum Corneum, that can be converted into arbitrary units of hydration. Corneometer measurement will be taken in the malar region of one randomized half of the face.
Number of Participants with Improvement From Baseline in Skin Appearance Assessed Using the Visia-CR Facial Imaging Booth | Baseline (Day 1), Day 7 and Day 28 +/- 2 days
  Facial images will be captured using the Visia CR Facial Imaging Booth. Three Three images per participant will be captured: right lateral, left lateral and frontal. The captured images will be further analyzed using specific image analysis software to evaluate improvement in the attributes of oiliness reduction, shine reduction, pore size reduction, and pore clearance, versus baseline and also between time-points.
Participant's Self-perceived Questionnaire to Assess the Clinical Effectiveness of the Sunscreen on Day 7 | Day 7
  Participant's self-perceived questionnaire to assess the clinical effectiveness of the sunscreen on Day 7 will be reported. Participants will answer 1 question on overall satisfaction with sunscreen by scoring as: disliked a lot, disliked, neither liked nor disliked, liked and liked a lot. Additionally, 15 attributes will be presented to be rated as: totally disagree, disagree, neither agree nor disagree, agree and totally agree.
Participant's Self-perceived Questionnaire to Assess the Clinical Effectiveness of the Sunscreen on Day 28 | Day 28
  Participant's self-perceived questionnaire to assess the clinical effectiveness of the sunscreen on Day 28 will be reported. Participants will answer 1 question on overall satisfaction with sunscreen by scoring as: disliked a lot, disliked, neither liked nor disliked, liked and liked a lot. Additionally, 15 attributes will be presented to be rated as: totally disagree, disagree, neither agree nor disagree, agree and totally agree.

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielli Brianezi, PhD, Principal Investigator — Johnson & Johnson Consumer Inc. (J&JCI)
Locations (1):
- Allergisa Pesquisa Dermato-Cosmética Ltda, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No